CLINICAL TRIAL: NCT06042907
Title: Development, Validation and Evaluation of the Feasibility of the Observational Risk Assessment of Contractures (Longitudinal Evaluation) Tool: The ORACLE Study
Status: Completed | Type: Observational
Sponsor: Bournemouth University (Other)
Collaborators: Dorset HealthCare University NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 45572
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Contracture; Joint Contracture
MeSH Terms: conditions — Contracture

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Observational Risk Assessment for Contractures- Longitudinal Evaluation (ORACLE) is a risk assessment tool for contractures. The tool was originally designed and developed by a group of multidisciplinary health professionals within Dorset Healthcare University NHS Foundation Trust (DHUFT). Bournemouth University and DHUFT sponsored a match funded studentship to establish the academic validation of the tool.

The results from the previously conducted studies (Phase One) as part of this project: (i) a systematic review of the literature and an (ii) online Delphi survey with field experts provided initial evidence for further development, content validity, and modification of the tool.

The current study (Phase Two) aims to establish the psychometric validation, acceptability, and usability of the modified tool through formal testing on adult care home residents in Dorset. It consists of two streams of work: Stream A aims to establish the psychometric validation by completing the ORACLE assessments on adult care home residents. The assessments will be performed by the care home staff. In Stream B, a realist evaluation will be performed to explore the usability and practicality of ORACLE with selected care home managers and staff who were involved in organising and completing the assessments on ORACLE respectively.

The results from this two-phase design will then inform further revisions of the tool if required.

DETAILED DESCRIPTION:
Joint contractures are described as any degree of reduction in the passive range of motion within a joint due to muscle or connective tissue shortening eventually leading to structural abnormalities within the affected joint. ). This can lead to further deterioration in limb and joint flexibility, mobility, and activities of daily living (ADL's).

It has been reported that the care home residents spend most of their time remaining sedentary. Reduced mobility or lack of physical activity adversely affects the residents' physical and psychological well-being of the residents, including reduced motivation to engage in physical and social activities, pain, increased risk of pressure sores, contractures, and physical dependency.

Structured risk assessments play an important role in referring patients to the appropriate health care practitioner and enacting early treatment strategies to reduce the risk of the condition progressing. However, there is a clear lack of a standardised, evidence-based measure that can actively identify the risk of contractures and trigger appropriate and timely referrals to healthcare professionals.

The tool, Observational Risk Assessment for Contractures- Longitudinal Evaluation (ORACLE) was initially designed with the aim to address the gap mentioned above by a group of healthcare professionals (physiotherapists, occupational therapists, and nurses within Dorset Healthcare, Bournemouth Borough Council, Poole Borough Council, Dorset County Council, and Dorset CCG. The working party discussed the potential causes and factors associated with contracture development and/or progression based on their clinical experience and developed relevant themes to define the construct of the tool. The original construct developed underwent a series of transformations before a face-to-face consensus over a series of meetings to finally include eight items in the tool.

To establish the academic validation of the tool before widespread use and implementation, Dorset Health Care collaborated with Bournemouth University and sponsored a match-funded PhD Studentship. The PhD project has been structured into two main phases: Phase One: content validation and phase II: external validation.

Phase One:

In the first phase, first a systematic review of literature was conducted collate evidence on factors associated with contractures in literature. Based on the findings of this review, an online two-round Delphi consensus survey was designed and conducted with a group of purposively sampled 30 panel experts to determine which items were significant for inclusion in ORACLE. The collective data provided by the systematic review and Delphi survey was then used to further develop and modify ORACLE.

Phase Two:

The current study (Phase Two) aims to establish the psychometric validation, acceptability, and usability of the modified tool through formal testing on adult care home residents in Dorset. It consists of two streams of work: Stream A aims to establish the psychometric validation by completing the ORACLE assessments on adult care home residents. The assessments will be performed by the care home staff. In Stream B, a realist evaluation will be performed to explore the acceptability and usability of ORACLE with selected care home managers and staff who were involved in organising and completing the assessments on ORACLE respectively. The results from this two-phase design will then inform further revisions of the tool if required.

ELIGIBILITY:
Inclusion Criteria:

• Care home residents aged 18 or above residing in residential and/ or nursing care homes located in Dorset.

Exclusion Criteria:

• Adults receiving end of life care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Care home residents will be recruited for this study
Sampling Method: Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Observational Risk Assessment for Contractures: Longitudinal Evaluation (ORACLE) | ORACLE (approx 10 minutes) will be administered thrice (twice by the same carer and once by a different carer) with a period of a 12-hour shift.
  The primary outcome measure in this study will be the newly developed contracture risk assessment tool (ORACLE) to evaluate its validity, reliability and acceptability in care homes

SECONDARY OUTCOMES:
Barthel Index | Barthel Index will be administered once (approx 10 minutes) in a 12 hour shift
  Barthel index is a standard measure of physical disability and assessment of performance in activities of daily living. This will be used to evaluate the convergent validity of ORACLE.

OTHER OUTCOMES:
Screening Questionnaire and Demographics | Screening questions and documents will be completed once within a 12 hour shift- approx 5 minutes
  A screening document will be completed to assess the eligibility of the residents.
  Non-identifiable demographics of the residents will also be recorded (e.g., age, gender, established contractures, co-morbidities etc).

CONTACTS AND LOCATIONS:
Overall Officials: Hina Tariq, Principal Investigator — Bournemouth University
Locations (8):
- United Kingdom (8):
  - Stratfield Lodge Care Home, Bournemouth, Dorset
  - Muscliff Nursing Home, Bournemouth, Dorset
  - Avon view, Christchurch, Dorset
  - Highcliffe Nursing Care Home, Christchurch, Dorset
  - Fernhill Dementia Home, Ferndown, Dorset
  - Branksome Park Care Centre, Poole, Dorset
  - Colten Care-Newstone House (Residential, Nursing and Dementia Care), Sturminster Newton, Dorset
  - Farway Grange Care Home, Bournemouth

REFERENCES:
- [Background] Bartoszek G, Fischer U, von Clarenau SC, Grill E, Mau W, Meyer G, Strobl R, Thiesemann R, Nadolny S, Muller M. Development of an International Classification of Functioning, Disability and Health (ICF)-based standard set to describe the impact of joint contractures on participation of older individuals in geriatric care settings. Arch Gerontol Geriatr. 2015 Jul-Aug;61(1):61-6. doi: 10.1016/j.archger.2015.03.005. Epub 2015 Mar 25. PMID 25937031
- [Background] Born CT, Gil JA, Goodman AD. Joint Contractures Resulting From Prolonged Immobilization: Etiology, Prevention, and Management. J Am Acad Orthop Surg. 2017 Feb;25(2):110-116. doi: 10.5435/JAAOS-D-15-00697. PMID 28027065
- [Background] Fergusson D, Hutton B, Drodge A. The epidemiology of major joint contractures: a systematic review of the literature. Clin Orthop Relat Res. 2007 Mar;456:22-9. doi: 10.1097/BLO.0b013e3180308456. PMID 17179779
- [Background] Forster A, Airlie J, Birch K, Cicero R, Cundill B, Ellwood A, Godfrey M, Graham L, Green J, Hulme C, Lawton R, McLellan V, McMaster N, Farrin A; REACH Programme Team. Research Exploring Physical Activity in Care Homes (REACH): study protocol for a randomised controlled trial. Trials. 2017 Apr 19;18(1):182. doi: 10.1186/s13063-017-1921-8. PMID 28424088
- [Background] Muller M, Fischer U, Bartoszek G, Grill E, Meyer G. Impact of joint contractures on functioning and social participation in older individuals--development of a standard set (JointConFunctionSet): study protocol. BMC Geriatr. 2013 Feb 21;13:18. doi: 10.1186/1471-2318-13-18. PMID 23432774
- [Background] Offenbacher M, Sauer S, Riess J, Muller M, Grill E, Daubner A, Randzio O, Kohls N, Herold-Majumdar A. Contractures with special reference in elderly: definition and risk factors - a systematic review with practical implications. Disabil Rehabil. 2014;36(7):529-38. doi: 10.3109/09638288.2013.800596. Epub 2013 Jun 17. PMID 23772994
- [Background] Skalsky AJ, McDonald CM. Prevention and management of limb contractures in neuromuscular diseases. Phys Med Rehabil Clin N Am. 2012 Aug;23(3):675-87. doi: 10.1016/j.pmr.2012.06.009. PMID 22938881
- [Background] Wagner LM, Clevenger C. Contractures in nursing home residents. J Am Med Dir Assoc. 2010 Feb;11(2):94-9. doi: 10.1016/j.jamda.2009.04.010. Epub 2010 Jan 15. PMID 20142063
- [Result] Tariq H, Collins K, Tait D, Dunn J, Altaf S, Porter S. Factors associated with joint contractures in adults: a systematic review with narrative synthesis. Disabil Rehabil. 2023 Jun;45(11):1755-1772. doi: 10.1080/09638288.2022.2071480. Epub 2022 May 11. PMID 35544581
- [Result] Tariq H, Collins K, Dunn J, Tait D, Porter S. The Delphi of ORACLE: An Expert Consensus Survey for the Development of the Observational Risk Assessment of Contractures (Longitudinal Evaluation). Clin Rehabil. 2024 May;38(5):664-677. doi: 10.1177/02692155241229285. Epub 2024 Feb 8. PMID 38332642